CLINICAL TRIAL: NCT06928701
Title: A Phase II Randomized Trial to Evaluate the Impact of "Targeted" Nutritional Apport and Exercise on the Modulation of Metabolic and Immune-related Gene Expression Signatures in Early Breast Cancer (eBC) Patients Candidate to Neoadjuvant Therapy (NAT)
Brief Title: Impact of "Targeted" Nutritional Apport and Exercise on the Modulation of Metabolic and Immune-related Gene Expression Signatures in Early Breast Cancer (eBC) Patients Candidate to Neoadjuvant Therapy (NAT)
Acronym: NEOMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Piedmont (Other)
Responsible Party: Principal Investigator, Alessandra Gennari, Principal Investigator, University of Eastern Piedmont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 02UPODIMETONCO
Record Dates: First submitted 2024-07-03; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Early Breast Cancer; Neoadjuvant Treatment
Keywords: treatment response; metabolomics; nutritional intervention
MeSH Terms: conditions — Breast Neoplasms | interventions — Docosahexaenoic Acids; Eicosapentaenoic Acid; hexadecenoic acid

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomised to one of 4 groups: A. NAT, according to molecular subtype; B. NAT plus nutritional supplementation; C. NAT plus supervised physical exercise; D. NAT plus supervised physical exercise plus nutritional supplementation. Nutritional supplementazion will consist of two main long-chain polyunsaturated fatty acids omega-3 (n-3 Lc-PUFA), EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) plus a source of palmitoleic acid (hexadecenoic acid).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A - treatment of physician choice (No Intervention): Conventional anti-cancer treatment, according to the molecular subtype and standard of care; all patients in Arm A will also receive general recommendations on lifestyle, including weight control and physical activity as indicated by WHO and EUSOMA criteria (control arm).
- B - nutritional supplementation (Experimental): Conventional anti-cancer treatment, according to the molecular subtype plus nutritional supplementation.
  Patients will be required to take on a daily basis two main long-chain polyunsaturated fatty acids omega-3 (n-3 Lc-PUFA), EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid), respectively at a dose of 700mg and 240mg, through 1 softgel twice a day. Besides, patients will be provided with a source of palmitoleic acid (hexadecenoic acid) equivalent to 1000mg of pure palmitoleic acid on a daily basis, through one daily 7 ml vial.
  Interventions: Dietary Supplement: omega-3 (n-3 Lc-PUFA), EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) plus a source of palmitoleic acid (hexadecenoic acid)
- C - physical activity (Experimental): Conventional anti-cancer treatment, according to the molecular subtype plus indication for supervised physical exercise
  Interventions: Dietary Supplement: omega-3 (n-3 Lc-PUFA), EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) plus a source of palmitoleic acid (hexadecenoic acid)
- D - nutritional supplementation plus physical activity (Experimental): Conventional anti-cancer treatment, according to the molecular subtype plus indication for supervised exercise training plus nutritional supplementation
  Interventions: Dietary Supplement: omega-3 (n-3 Lc-PUFA), EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) plus a source of palmitoleic acid (hexadecenoic acid)

INTERVENTIONS:
Dietary Supplement: omega-3 (n-3 Lc-PUFA), EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) plus a source of palmitoleic acid (hexadecenoic acid) — Nutritional supplements
  Arms: B - nutritional supplementation; C - physical activity; D - nutritional supplementation plus physical activity

SUMMARY:
NEOMET is an exploratory randomized prospective, multicenter study whose primary aim is to explore if metabolomic signatures can be modified by a lifestyle intervention including dietary supplements and physical exercise intervention, in eBC patients candidate to NAT. Eligible patients will be randomised to one of 4 groups: A. NAT, according to molecular subtype; B. NAT plus nutritional supplementation; C. NAT plus supervised physical exercise; D. NAT plus supervised physical exercise plus nutritional supplementation. Nutritional supplementazion will consist of two main long-chain polyunsaturated fatty acids omega-3 (n-3 Lc-PUFA), EPA (eicosapentaenoic acid) and DHA (docosahexaenoic acid) plus a source of palmitoleic acid (hexadecenoic acid).

DETAILED DESCRIPTION:
The primary objectives are: 1. To explore the impact of a lifestyle intervention including dietary supplements and physical exercise on the modulation of metabolomic signatures in eBC patients candidate to NAT; 2. To assess the Omega-3 Index at baseline and before surgery in all patient cohorts. Secondary objectives are: Impact of the combined lifestyle intervention on patient metabolic profile and body composition, by bioelectrical Impedance analysis; assessment of the immunophenotype of lymphocyte subpopulations and their correlation with metabolomic profile and response to therapy; characterization of immune-related and metabolic-related gene-expression signatures in tumor tissue and their correlation with metabolomic profile and response to therapy; evaluation of the pharmacokinetic interactions between nutritional supplementation and chemotherapy; evaluation of pCR in the different treatment arms; changes in health-related QoL (EORTC QLQ-C30, QLQ-BR45, and EQ-5D-5L), and safety and toxicity profiles according to the NCI-CTCAE v.5.0.

Due to explorative intent of the study no formal sample size calculation is provided. A total of 160 consecutive patients will be enrolled into the four arms of the study, with an allocation ratio equal to 1:1:1:1 (40 pts/arm). It can be estimated that the accrual will be completed in 20 months. Data collection, molecular assessments and data analysis with final scientific output are expected to extend the study duration to a total of 26 months.

The following analyses will be performed: - Conversion rate from a poor to a good metabolomic prognostic signature from baseline to end of NAT. - Change in Omega-3 Index and body composition variation.

- The association between Immunophenotype of lymphocyte subpopulations and tissue-based metabolic and immune-related gene-expression signatures will be described according to the type of metabolomic profile at baseline (poor versus good) and with response to therapy (pCR versus RD).

ELIGIBILITY:
Inclusion Criteria:

* - Women (regardless of menopausal status) ≥ 18 years of age
* Pathologic confirmation of breast cancer by tumor biopsy
* Immunohistochemical assessment (as per local standards) of ER and PgR status, HER2 status;
* Stage I-III breast cancer without evidence of distant metastases
* Being candidate to standard neoadjuvant therapy
* Having available tumor tissue from breast and/or lymph node at baseline
* Ability to fill a nutritional daily diary
* Medical clearance for non-agonistic physical activity
* Written informed consent to study-specific procedures

Exclusion Criteria:

* - locally advanced or inflammatory or stage IV BC;
* tumor size < 1 cm with negative nodes (pT1a, N0);
* chronic diseases or orthopedic issues that might interfere with ability to undertake a dietary and physical activity program;
* personal history of eating disorders.
* women engaged in agonistic/vigorous sport activities, not able to be compliant to exercise schedules

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Variation of fatty acids concentration | T0: baseline, prior to cycle 1 (each cycle is 21 days); T1: end of NACT, before surgery (NACT is approximately 6 months, according to biological subtype)
  Plasma metabolic sample will be analyzed using a GCxGC-MS instrument for the relative and absolute quantification of small molecules in order to evaluate the impact of a lifestyle intervention including dietary supplements and physical exercise on the modulation of metabolomic signatures in eBC patients candidate to NACT.
Omega3 Index | T0: baseline, prior to cycle 1 (each cycle is 21 days); T1: end of NACT, before surgery (NACT is approximately 6 months, according to biological subtype)
  Assessment of Omega-3 Index in all patients cohorts at:
  * baseline
  * pre-operatative (at the end of NACT)
  The omega3 index will assessed by the sum of DHA and EPA in erythrocytes expressed as a percentage of total erythrocyte fatty acid.

SECONDARY OUTCOMES:
Combined lifestyle intervention | T0: baseline, prior to cycle 1 (each cycle is 21 days); T1: end of NACT, before surgery (NACT is approximately 6 months, according to biological subtype)
  Impact of the combined lifestyle intervention on body composition. Body composition will be assessed with a multifrequency bioelectrical impedance analysis.
Lymphocyte subpopulations | T0: baseline, prior to cycle 1 (each cycle is 21 days); T1: end of NACT, before surgery (NACT is approximately 6 months, according to biological subtype)
  Assessment of the immunophenotype of lymphocyte subpopulations and their correlation with metabolomic profile and response to therapy; characterization of immune-related and metabolic-related gene-expression signatures in tumor tissue and their correlation with metabolomic profile and response to therapy.
  Lymphocyte subpopulation will be assessed collecting blood at 1st cycle and at the last cycle of NACT (before surgery). Gene-expression signatures will be assessed on tumor biopsy and surgery tissue.
Antitumor activity | From T0 until surgery, approximately 6 months (according to biological subtype)
  evaluation of pathological Complete Response (pCR) in the different treatment arms (ypT0/Tis ypN0)
changes in health-related Quality of Life | T0: baseline, prior to cycle 1 (each cycle is 21 days); T1: at three months after inclusion; T2: end of NACT, before surgery (NACT is approximately 6 months, according to biological subtype)
  Quality of Life will be assessed among all patients included in the study using patient-reported outcomes (PROs) collected using a validated and standardized questionnaire: the European Organization for Cancer Research and Treatment Quality of Life Questionnaire C30, ranging from 0 to 100. A high-scale score represents a higher response level.
changes in health-related Quality of Life | T0: baseline, prior to cycle 1 (each cycle is 21 days); T1: at three months after inclusion; T2: end of NACT, before surgery (NACT is approximately 6 months, according to biological subtype)
  Quality of Life will be assessed among all patients included in the study using patient-reported outcomes (PROs) collected using a validated and standardized questionnaire: the European Organization for Cancer Research and Treatment Quality of Life Questionnaire BR45, ranging from 0 to 100. A high-scale score represents a higher response level.
changes in health-related Quality of Life | T0: baseline, prior to cycle 1 (each cycle is 21 days); T1: at three months after inclusion; T2: end of NACT, before surgery (NACT is approximately 6 months, according to biological subtype)
  Quality of Life will be assessed among all patients included in the study using patient-reported outcomes (PROs) collected using a validated and standardized questionnaire: Hospital Anxiety and Depression Scale, ranging from 0 to 21. A high-scale score represents a lower response level (0-7 normal, 8-10 borderline, 11-21 abnormal).
Impact on treatment-related adverse events | Evaluation will be performed before of each cycle of NACT (each cycle is 21 days). NACT is approximately 6 months, according to biological subtype.
  Evaluation of safety and toxicity profiles according to the NCI-CTCAE (Common Terminology Criteria for Adverse Events) v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Gennari, MD, Study Chair — University of Piemonte Orientale
Locations (1):
- AOU Maggiore della Carità, Novara, Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided